CLINICAL TRIAL: NCT02993419
Title: Bacillus Particles Prevent More Children's Antibiotic-associated Diarrhea (AAD), Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Bacillus Particles Prevent Children Antibiotics Associated Diarrhea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dbzy160801
Record Dates: First submitted 2016-08-18; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bacillus licheniformis Intervention (Experimental): The intervention is use Bacillus licheniformis particles，The drugs 1 bag each time, three times a day, for taking seven days; children observed during the test is no longer taking other probiotic preparations, and any other proprietary Chinese medicine preparation
  Interventions: Drug: Bacillus licheniformis Intervention
- placebo Intervention (Placebo Comparator): The intervention is use placebo，The drugs 1 bag each time, three times a day, for taking seven days; children observed during the test is no longer taking other probiotic preparations, and any other proprietary Chinese medicine preparation
  Interventions: Other: placebo Intervention

INTERVENTIONS:
Drug: Bacillus licheniformis Intervention — On the basis of the use of antibiotics in children with symptomatic treatment, the addition of experimental drugs 1 bag each time, three times a day, for taking seven days; children observed during the test is no longer taking other probiotic preparations, and any other proprietary Chinese medicine preparation
  Arms: Bacillus licheniformis Intervention
Other: placebo Intervention — On the basis of the use of antibiotics in children with symptomatic treatment, the addition of placebo drugs 1 bag each time, three times a day, for taking seven days; children observed during the test is no longer taking other probiotic preparations, and any other proprietary Chinese medicine preparation
  Arms: placebo Intervention

SUMMARY:
This prospective, multicenter, randomized, double-blind, placebo-controlled clinical study, into the group of children in the hospital that use clinical antibiotics from one month to three years old，by observing the given antibiotics at the same time with the whole bowel raw or placebo, prevent the happening of the antibiotic associated diarrhea, evaluate the whole bowel prevention clinical efficacy and safety of AAD.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized, double-blind, placebo-controlled clinical study, into the group of children in the hospital that use clinical antibiotics from one month to three years old，by observing the given antibiotics at the same time with the whole bowel raw or placebo, prevent the happening of the antibiotic associated diarrhea, evaluate the whole bowel prevention clinical efficacy and safety of AAD.

Outcome measures

1. MAIN OUTCOME MEASURES: The incidence of diarrhea (stool frequency and character daily rates), the duration of diarrhea, the degree of diarrhea occur.
2. Secondary outcomes: intestinal flora and relevant metabolites, micro-environmental changes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1-3 years
2. no diarrhea-related symptoms
3. the diagnosis of lower respiratory tract infection (acute bronchitis, pneumonia) in hospitalized children
4. the need for penicillins, cephalosporin antibiotic treatment, treatment for 7-14 days, combined with other antimicrobial agents alone
5. parent or guardian signed informed consent (6）Not used in children with related traditional Chinese medicine injection

Exclusion Criteria:

1. diarrhea in the group, or 2 weeks before admission into children with diarrhea
2. children with ICU wards, digestive tract malformations, children with gastrointestinal surgery, congenital heart disease, artificial heart surgery, children with rheumatic heart disease, infective endocarditis
3. receiving immunosuppressive agents in children
4. Children who received any probiotic preparation 2 weeks before enrollment

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-09 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Record daily stool frequency, shape observation excrement | every day，A total of seven days
  Record daily stool frequency, excrement shape. According to Bristol who Chart of shape evaluation standard of excrement and urine, feces traits can be divided into seven grades, as picture shown in feces traits scale, record with feces corresponding score, score 5 or more, it indicates that the waste is not normal, diarrhea symptoms

SECONDARY OUTCOMES:
Strain type | the first day and the seven day
  Detection of intestinal strains of the species

IPD SHARING:
Plan to Share IPD: Undecided